CLINICAL TRIAL: NCT02272881
Title: The Santa Barbara Pressure Ulcer Study Comparison of Immediate Flap Closure Versus Wound Care for Management of Late-stage Pressure Ulcers: a Randomized, Prospective Clinical Trial
Brief Title: A Randomized, Prospective Clinical Trial of Immediate Flap Closure Versus Wound Care for Management of Late-stage Pressure Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have not been able to enroll patients.
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-42r
Record Dates: First submitted 2014-10-09; First posted 2014-10-23 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate surgical intervention (Experimental): immediate surgical reconstruction of the pressure ulcer via flap closure or comparable procedure
  Interventions: Procedure: surgical reconstruction
- wound care (Other): conservative wound management directed by certified wound care experts
  Interventions: Procedure: wound management

INTERVENTIONS:
Procedure: surgical reconstruction — Patients randomized to surgical flap closure will undergo reconstructive plastic surgery to close an intended pressure ulcer at the earliest date after selection. Our group's co-investigator and staff plastic and reconstructive surgeon will decide on the optimal technical repair. Given the lack of retrospective evidence to support a superior surgical repair (myocutaneous, fasciocutaneous, local flap arrangement versus free microvascular tissue transfer) we will defer to our physician staff preference on a per patient basis. The time from enrollment to surgical intervention will be tracked, and no patient will be dropped from the study should this time exceed the two-week ideal.
  Arms: immediate surgical intervention
Procedure: wound management — Patients selected to the supportive wound care arm will be managed by the Center for Wound Care at Cottage Health System, a certified wound care center. They will receive standard of care conservative wound care including: debridement, dressing changes, wound checks, physical therapy, occupational therapy, antibiotic treatment, nutritional support and close follow-up over the study period.
  Arms: wound care

SUMMARY:
The purpose of this study is to compare the number of and degree of pressure ulcers healed, as measured by intact skin at the original ulcer site at 6 months of follow-up in patients randomized to immediate operative closure versus those who are maintained in a wound care program in patients with Stage 3 and 4 sacral and peri-sacral decubitus ulcers.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Stage III or IV pressure ulcers on or near trochanter, ischium, sacrum or buttocks;
* Receiving treatment at the Center for Wound Management - Goleta Valley Cottage Hospital; Santa Barbara Cottage Hospital or Santa Ynez Cottage Hospital, all part of Cottage Health System;
* Underlying etiology for immobility secondary to spinal cord injury (SCI) or other neuromuscular condition not expected to become progressive in next 12 months;
* No contraindications to undergo surgical intervention, including medical ability to tolerate surgical procedure with general anesthesia.

Exclusion Criteria:

* Unable or unwilling to provide informed consent;
* Underlying cause of immobility secondary to chronic medical disease outside of nonprogressive SCI or neuromuscular disease as described above;
* Patients requiring immediate surgical closure determined by physician judgment;
* Those deemed inappropriate to consider for surgery outside of study; potential reasons normally include medical comorbidities, inability to comply with post-operative care, and lack of funding source for elective procedure, peri-operative, and / or wound care.
* Patients who have already been receiving active, professionally supervised wound care for > 2 week period prior to presentation
* Patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 6 months after randomization
  measured by intact skin at the original ulcer site